CLINICAL TRIAL: NCT01935063
Title: A Comparison of Cognitive-behavioral Couple Therapy and Lidocaine in the Treatment of Provoked Vestibulodynia: A Randomized Clinical Trial
Brief Title: Study to Compare the Efficacy of Cognitive-behavioral Couple Therapy and Lidocaine for Provoked Vestibulodynia
Acronym: CBCT-RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Responsible Party: Principal Investigator, Sophie Bergeron, Associate Professor, Psychology, Université de Montréal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBCT-02; 299610 (Other Grant/Funding Number: Canadian Institutes of Health Research (CIHR))
Record Dates: First submitted 2013-08-27; First posted 2013-09-04 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Vulvodynia; Dyspareunia; Vestibulodynia
Keywords: Vulvodynia; Provoked vestibulodynia; Vulvar pain; Dyspareunia; Couples therapy; Lidocaine; Cognitive behavioral couple therapy; Cognitive behavioral therapy; Pain; Pain during sexual intercourse
MeSH Terms: conditions — Vulvodynia; Dyspareunia; Pain | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive Behavioral Couple Therapy (Experimental): CBCT is a 12-session therapy that includes the following: re-conceptualize PVD as a multidimensional pain problem influenced by a variety of factors including thoughts, emotions, behaviours and couple interactions; psychoeducation about PVD and its impact upon sexuality, defining/working the sexual script, mindfulness techniques, communication skills training, and sexual approach/avoidance goals work, defusion and acceptance approaches to coping with pain, among others.
  Interventions: Behavioral: Cognitive Behavioral Couple Therapy
- Topical lidocaine (Active Comparator): Nightly applications of a 5% lidocaine ointment on the vulvar vestibule, at the entry of the vagina (50mg/g, Xylocaïne®, AstraZeneca, tube of 35g) for 12 weeks, as described by Zolnoun et al. (Zolnoun, Hartmann, & Steege, 2003).
  Interventions: Other: Topical Lidocaine

INTERVENTIONS:
Behavioral: Cognitive Behavioral Couple Therapy — CBCT includes the following: (1) re-conceptualize PVD as a multidimensional pain problem influenced by a variety of factors including thoughts, emotions, behaviors and couple interactions; (2) re-conceptualize PVD as a couple problem in which both members of the couple affect and are affected by the pain; (3) modify those factors associated with pain during intercourse with a view to increasing adaptive coping, for example, by increasing self-efficacy and decreasing catastrophizing, as well as decreasing pain intensity; (4) improve the quality of sexual functioning, reduce sexual distress and increase sexual satisfaction; (5) consolidate skills.
  Other Names: CBCT
  Arms: Cognitive Behavioral Couple Therapy
Other: Topical Lidocaine — Nightly applications of a 5% lidocaine ointment on the vulvar vestibule, at the entry of the vagina (50mg/g, Xylocaïne®, AstraZeneca, tube of 35g) for 12 weeks, as described by Zolnoun et al. (2003). In addition, the cream will be applied to a cotton ball kept on the vestibule via the participant's underwear overnight to ensure a continued 7 to 8-hour contact between the anesthetic and the vestibule. A pamphlet with figures detailing how to apply the cream will be given to participants, in addition to a calibrated measurement tool to ensure that all participants apply the same quantity every night.
  Other Names: Lidocaine; Xylocaine (R); Nightly lidocaine
  Arms: Topical lidocaine

SUMMARY:
Chronic pain problems involving the female reproductive system are major health concerns for all women. Poorly understood, they entail great personal and financial cost. One such condition is vulvodynia, or chronic unexplained vulvar pain, which has a prevalence of 16%. Despite its negative impact on psychosexual and relationship satisfaction, there is little research examining empirically-tested treatments for afflicted couples. The proposed research builds on findings from our work focusing on the impact of relational factors on vulvodynia, and our previous research evaluating the efficacy of group cognitive-behavioral therapy for this problem. This two-centre randomized clinical trial aims to assess the efficacy of a novel, 12-week targeted couple therapy (CBCT) for women with vulvodynia in comparison to one of the most commonly prescribed first line medical interventions, topical lidocaine. Primary research question: Is there a significant difference between the two treatments on women's pain during intercourse post-treatment? Secondary research questions will assess for significant differences between the two treatments post-treatment and at 6-month follow-up on multidimensional aspects of pain using the McGill Pain Questionnaire, women and partners' sexuality (sexual function and satisfaction), psychological adjustment (anxiety, depression, catastrophizing, self-efficacy, attributions, and quality of life), relationship factors (partner responses, couple satisfaction, attachment, and communication styles), and self-reported improvement and treatment satisfaction. Results of this study will improve the health and quality of life of patients with vulvodynia by rigorously testing the efficacy of a novel couples treatment.

DETAILED DESCRIPTION:
Background: Chronic pain problems involving the female reproductive system are major health concerns in women of all ages. As conditions which are poorly understood and often misdiagnosed or ignored, they entail a great personal cost to patients and a significant financial cost to society. One such condition is vulvodynia, or chronic unexplained vulvar pain. A recent population-based study suggests that the lifetime cumulative incidence of vulvodynia is 16%, indicating that approximately 2.5 million Canadian women may experience idiopathic vulvar pain during their lifetimes. Provoked vestibulodynia (PVD) - an acute recurrent pain localized within the vulvar vestibule and experienced primarily during sexual intercourse - is suspected to be the most frequent cause of vulvodynia in premenopausal women, with prevalence estimates of 12% in community samples. Despite its high prevalence and negative impact on psychosexual functioning, there has been a paucity of controlled research to provide empirically validated treatments for afflicted couples. The present proposal draws on our previous cross-sectional and prospective CIHR funded research on the dyadic determinants of pain and psychosexual impairment in women with PVD and their partners, as well as on our past randomized trials evaluating the efficacy of group cognitive-behavioral therapy for this condition. Specifically, the goal of our study is to evaluate the efficacy of a targeted cognitive-behavioral couple therapy (CBCT) intervention that we developed for the treatment of PVD.

Objectives: The proposed two-centre randomized clinical trial aims to evaluate the efficacy of a novel 12-week targeted couple therapy intervention (CBCT) for women with PVD in comparison to one of the most frequently prescribed first line medical interventions, topical lidocaine, shown to be effective and safe in the management of PVD. The primary research question focuses on whether there is a significant difference between the two treatments on women's pain during intercourse post-treatment. Secondary research questions focus on whether there are significant differences between the two treatments post-treatment and at 6-month follow-up on (a) the multidimensional aspects of women's pain on the McGill Pain Questionnaire and (b) women and partners' sexuality (sexual function and satisfaction, frequency of intercourse), psychological adjustment (anxiety, depression, catastrophizing, self-efficacy, pain attributions, quality of life, acceptance of pain, compassionate love for partner, self-compassion, emotion regulation and thoughts and feelings related to pain experience), relationship factors (partner responses, dyadic adjustment, attachment, and communication) and self-reported improvement and treatment satisfaction. We will also examine whether childhood trauma and co-morbid pain conditions moderate treatment response. Finally, a third research question is to evaluate the role of hormonal contraceptive use and the risk of PVD.

Research plan/methodology: The proposed research is a 3.5-year, two-centre parallel randomized controlled trial for PVD using an intent-to-treat analysis strategy, with pain during intercourse as the primary outcome. The main research questions will be addressed by: 1) recruiting 224 premenopausal women and their partners with medically diagnosed PVD; 2) performing comprehensive gynecological and psychosexual pre-treatment evaluations focusing on our outcome measures; 3) randomly assigning women to one of the two 12-week treatment arms: CBCT or lidocaine, and 4) evaluating pain during intercourse, as well as sexual, psychological and relationship outcomes, in addition to self-reported improvement and treatment satisfaction, post-treatment and at 6-month follow-up. These procedures will take place in two different university centers: Université de Montréal in Montréal, Québec, and Dalhousie University in Halifax, Nova Scotia, and their affiliated hospitals. Both university centres will store data securely, adhering to the protocols outlined by the ethics review boards at each site.

Statistical Analyses: Analyses will be conducted based on intention to treat. Descriptive statistics will be used to define and compare the participants in both intervention groups. More specifically, we will calculate means, medians, deviations and interquartile ranges and T-tests will be used to determine the differences between groups for socio-demographic variables. Chi-square tests and observed differences between groups will be used for categorical variables. If differences are observed between groups, these variables will be controlled for in subsequent analyses. We will verify that variables are normally distributed. If variables are not normally distributed, non-parametric tests will be employed. A repeated measures analysis of variance will permit the assessment of efficacy of the two treatments at post-treatment and at 6-month follow-up. The analyses will focus on the changes in pain experienced during intercourse from pre-treatment assessment to post-treatment and 6-months follow-up. To do this, time will be the intra-subject variable, and the experimental condition will be the inter-subject variable.

For secondary analysis, multiple analyses will be conducted in multiple steps, with multivariate analyses being conducted first for repeated measures (MANOVA). Correlated measures will be grouped based on conceptual domain (e.g., pain, dyadic adjustment, catastrophizing). Univariate analyses will be conducted if the multivariate results are significant (ANOVA). This will be followed by orthogonal contrasts to examine changes between different measurements. Moreover, we will use exploratory analyses for participants who completed the experimental protocol to determine the effect protocol adherence has on treatment efficacy. Multiple regression analyses will be used to examine the link between socio-demographic variables, pre-treatment dependent variables and pain at post-treatment and 6-months follow-up to identify factors associated with therapeutic success. These latter analyses will be conducted for each treatment group separately. Bonferroni corrections will be used during analyses for multiple comparison adjustments. In the case of missing data, we will explore the effects of withdrawal on sensitivity analyses, replace the missing data with data from the most recent assessment or with averaged or aggregate values.

Significance of study: Results of the proposed research may improve the health and quality of life of Canadians afflicted with a highly prevalent and neglected women's health problem - vulvodynia - by providing a rigorous test of the efficacy of a novel targeted couple therapy intervention.

ELIGIBILITY:
Inclusion Criteria:

* pain during intercourse which a) is subjectively distressing, b) occurs on 80% of intercourse attempts, and c) has lasted for at least six months;
* pain limited to intercourse and other activities involving pressure to the vestibule;
* ability to undergo the gynecological examination to completion;
* significant pain in one or more locations of the vestibule during the gynecological exam, which is operationalized as a minimum patient pain rating of 4 on a scale of 0 to 10;
* having engaged in vaginal intercourse as a couple once per month for the last three month;
* partnered in a committed, monogamous relationship for at least 6 months; and
* has had at least four in-person contacts per week with their partner for at least six months.
* Partners will be recruited conditional upon the patient meeting study selection criteria.
* Both women and partners must be able to read, speak, and understand English or French (in Montreal), and English (in Halifax) to participate.

Exclusion Criteria:

* vulvar pain not clearly linked to intercourse or pressure applied to the vestibule;
* presence of one of the following: a) major medical and/or psychiatric illness, b) active infection, c) dermatologic lesion, d) pregnancy or planning a pregnancy;
* age less than 18 for couples or greater than 45 for women with pain;
* major medical and/or psychiatric illness for partners;
* severe relational distress or conflict as determined by baseline measures and interview;
* current participation in another couple therapy, or therapy/treatment related to PVD.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2014-03-06 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-12-10 (Actual)

PRIMARY OUTCOMES:
Change in pain during intercourse / sexual activity from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Pain during intercourse will be assessed using a visual analog scale (VAS) ranging from 0 to 10, where 0 is no pain at all, and 10 is the worst pain ever, as recommended by the IMMPACT guidelines for chronic pain clinical trials (Dworkin et al., 2005). Participants will report on pain experienced in the preceding month. The main outcome will be the change in the VAS scores from pre- to post-treatment. This measure has been shown to detect significant treatment effects in women with PVD (Bergeron et al., 2001) and demonstrates a significant positive correlation with other pain intensity measures. Pain during intercourse is the main symptom of PVD and the one that most interferes with quality of life, hence the most relevant measure of functional outcome.

SECONDARY OUTCOMES:
Change in qualitative components of pain from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Qualitative components of pain will also be assessed using the Short-Form McGill Pain Questionnaire (MPQ; Melzack, 1985), a measure of the sensory, affective and evaluative components of pain. The MPQ is a widely used adjective 15-item checklist which assesses both qualitative and quantitative aspects of pain (Grafton, Foster, & Wright, 2005; Melzack & Katz, 2001). We will use the Pain Rating Index (PRI) scale.
Changes in partner responses to pain from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Partner responses from the point of view of the women with PVD and their partners will be measured with the West Haven-Yale Multidimensional Pain Inventory - Significant Other Response Scale (MPI; Kerns, Turk, & Rudy, 1985), and the Spouse Response Inventory - Facilitative subscale (SRI; Schwartz, Jensen, & Romano, 2005) which have been adapted to our PVD population and their partners.
Change in dyadic adjustment from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Dyadic adjustment will be assessed using the Couple Satisfaction Index (CSI; Funk & Rogge, 2007), a 32-item measure of relationship satisfaction. Compared to other well-known relationship satisfaction measures (e.g., Dyadic Adjustment Scale; Spanier, 1976) it demonstrates strong convergent validity, and a higher precision and power for detecting distinctions in satisfaction levels (Funk & Rogge, 2007). Moreover, unlike similar relationship satisfaction scales, the CSI has been tested with a sample of participants spanning the relationship spectrum (e.g., dating, engaged, married).
Change in pain catastrophizing for both women and partners from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale (PCS; Sullivan, Bishop, & Pivik, 1995), which consists of 13 items scored on a 5-point scale with the end points (0) not at all and (4) all the time. The PCS is divided into three subscales: rumination, magnification and helplessness. It is a reliable and valid measure that has demonstrated a stable factorial structure across clinical and general populations, including a French population (Sullivan, Bishop, & Pivik, 1995; Osman et al., 2000; French et al., 2005). Cano et al. (Cano, Leonard, & Franz, 2005) recently validated a partner version and found excellent psychometric properties.
Changes in pain attributions from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Pain attributions will be measured with the Extended Attributional Style Questionnaire (EASQ; Metalsky, Halberstadt, & Abramson, 1987), adapted for use with women who experience genital pain, and their partners. The adapted EASQ consists of 12 hypothetical negative situations that occur within a genital pain context, and participants are asked to indicate the major cause of the situation (open-ended), and then rate the cause on the following dimensions: internal, global, and stable on a 7-point Likert scale. The EASQ adapted for genital pain demonstrates good internal consistency (alpha=0.84-0.86) for subscales and total score, as well as a similar factor structure to the original EASQ (Jodoin et al., 2011). We have used both the woman and partner version successfully in previous studies (Jodoin et al., 2008; 2011).
Change in anxiety from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Both partners will complete the Trait Anxiety subscale of the Spielberger State-Trait Anxiety Inventory (STAI - (Spielberger, Gorsuch, & Lushene, 1970). This 20-item, well-known, and widely used measure has demonstrated very good psychometric properties in clinical and non-clinical populations, including in chronic pain (Gauthier & Bouchard, 1993; Greenberg & Burns, 2003; Rule & Traver, 1983; Tanaka-Masumi & Kameoka, 1986).
Change in depression symptoms to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Both partners will complete the Beck Depression Inventory-Fast Screen (BDI-FS; Beck, Steer, & Brown, 1996; Beck, Steer, & Garvin, 1988), an adapted 7-item version of the widely-used 21-item measure. Specifically, the BDI-FS assesses sadness, loss of pleasure (anhedonia), suicide ideation, pessimism, past failure, self-dislike and self criticalness with scores for items ranging from 0 (low intensity) to 3 (high intensity). This measure has been used with chronic pain populations (Poole, Bramwell, & Murphy, 2008).
Change in pain self-efficacy of women with PVD from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Pain self-efficacy will be assessed using the Painful Intercourse Self-Efficacy Scale (PISES; Desrochers et al., 2009), which was adapted from the Arthritis Self-Efficacy Scale (Lorig et al., 1989). The PISES consists of 20 items with three subscales: self-efficacy for controlling pain during intercourse, for sexual function, and for other symptoms. Participants indicate their perceived ability to carry out sexual activity or to achieve outcomes in pain management by responding on a scale from 10 (very uncertain) to 100 (very certain). Higher scores indicate greater self-efficacy. The reliability and validity of the original version have been established (Lorig et al., 1989) and the factor structure of the adapted version has been shown to be identical to that of the original (Desrochers, 2009). In our previous samples, Cronbach's alphas ranged from .79 to .89 for women and .74 to .91 for partners.
Self-reported improvement following treatment (duration of treatment is 12 weeks) | Post-treatment, and 6-months post-treatment
  Woman and partner self-reported improvement [scale of 0 (worse) to 5 (complete cure)] and treatment satisfaction [scale of 0 (completely dissatisfied) to 10 (completely satisfied)] will be measured post-treatment and at 6-month follow-up to assess the clinical significance of results.
Change in sexual satisfaction for both partners from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Sexual satisfaction will be assessed using the Global Measure of Sexual Satisfaction scale, which consists of 5 items assessing global sexual satisfaction. Internal consistency of this scale is high (alpha = 0.90), as is test-retest reliability (r = 0.84; Lawrence & Byers, 1998).
Changes in sexual function from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Sexual function for both women and their partners will be assessed using the Derogatis Interview for Sexual Functioning - Self-Report (DISF-SR), a 25-item self-report measure of sexual function for men and women (Derogatis, 1997). It covers five dimensions of sexuality: sexual cognition/fantasy, arousal, sexual behaviour/experience, orgasm, and sexual drive/relationship. Scores can be calculated for each dimension and for global sexual functioning. The DISF-SR boasts good internal consistency and reliability (Derogatis, 1997; Meston & Derogatis, 2002; Daker-White, 2002).
Changes in quality of life from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Both partners will complete the Quality Metric™ Short Form 12-question Health Survey (SF-12). This reliable and valid survey was adapted from the widely-used SF-36 health survey and assesses physical and mental health and wellness across 8 scales: physical function, bodily pain, vitality, general health, emotional and physical roles, social functioning, and mental health (Cheak-Zamora, Wyrwich, & McBride, 2009; Ware, Kosinski, Keller, 1996). The SF-36 has been used previously in PVD samples (Sutton, Pukall, & Chamberlain, 2009).
Changes in attachment, or experiences in close relationships from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Attachment will be measured using the Experiences in Close Relationships Scale-Revised (ECR-RS; Wei, Russel, Mallinckrodt, & Vogel, 2007). The ECR-RS is a 12-item scale that assesses components of adult attachment (e.g., secure, anxious, avoidant attachment). Both members of the couple will complete this measure.
Change in interpersonal sexual goals from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Approach and avoidance interpersonal sexual goals will be assessed with a 15-item measure adapted from Cooper et al. (1998) (Impett, Peplau, & Gable, 2005; Impett et al., 2008; Impett, Gordon, & Strachman, 2008). Participants rate the importance of 9 approach and 6 avoidance interpersonal goals in influencing their decision to engage in sex on a 7-point scale. This measure has demonstrated high internal consistency (Impett et al., 2005; Impett et al., 2008).
Changes in communication patterns from baseline, and over the course of treatment | Baseline, Weeks 1, 4, 8, and 12 of treatment
  At the pre-treatment, post-treatment, and follow-up evaluation sessions, both partners will complete the Communication Patterns Questionnaire - Short Form (Christensen & Heavey, 1990), an 11-item measure of communication patterns during couples' discussions of problems. This measure examines three overall patterns of communication: conflict avoiding, conflict engaging, and positive interaction (Futris et al., 2010). This measure has demonstrated good psychometric properties (Futris, Campbell, Nielsen, & Burwell, 2010). We will also collect 12 additional items from the full measure to assess the subscales of mutual avoidance, mutually constructive communication, and other communication patterns during and after periods of conflict (Christensen & Shenk, 1991).
Change in intimacy ratings from baseline, and over the course of treatment | Baseline, Weeks 1, 4, 8, and 12 of treatment
  Both partners will complete measures of general relationship intimacy (8-items; Laurenceau et al., 2005) and sexual intimacy (12-items; Bois et al., 2013). These measures assess self-disclosure, partner disclosure, and partner responsiveness in the context of the interpersonal exchanges and sexual activity. They have demonstrated high internal consistency in our previous PVD research (Bois et al., 2013).
Changes in Fear of Pain from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Fear of pain will be measured using the Pain Anxiety Symptoms Scale (PASS-20; McCracken & Dhinga, 2002), a 20-item, self-report measure of fear of pain designed for individuals with chronic pain problems and has been adapted for use in a sexual context (i.e. the word sexual has been added before the word activity for several items). Subscales include: Cognitive Anxiety, Escape/Avoidance, Fearful appraisal, and Physiological Anxiety. Only women with PVD will complete this measure.
Changes in Hypervigilance to Pain from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Hypervigilance to pain during intercourse will be assessed with the Pain and Vigilance Awareness Questionnaire (PVAQ); McCracken, 1997), a 16-item measure of attention to pain that has been used to evaluate awareness, consciousness and vigilance to pain in various clinical and non-clinical populations. It shows good test-retest reliability and internal consistency (Roelofs et al., 2003). Only women with PVD will complete this measure.
Changes in Acceptance of Chronic Pain from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Both partners will complete an adapted version of the Chronic Pain Acceptance Questionnaire (McCracken, Vowles, &Eccleston, 2004) for use with women experiencing vulvovaginal pain and their partners. This 20-item scale measures acceptance and openness to experiencing pain sensations, and the pursuit of a satisfying life in spite of pain. The partner version references their own acceptance of their partner's pain. A recent systematic review of measures of acceptance of chronic pain indicated that, based on psychometric properties, there is the most support for use of the CPAQ to measure acceptance of pain in chronic pain patients, as compared to other questionnaires (Reneman et al., 2010). Studies using the CPAQ have found Cronbach's alpha of the sum score that ranges from 0.78-0.85.
Changes in female sexual function from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Only women with PVD will complete the Female Sexual Function Inventory (FSFI), a self-report 19-item measure assessing sexual functioning in women such as sexual arousal, orgasm, sexual satisfaction and discomfort experienced during sexual activity and intercourse with high internal consistency (i.e., high inter-item correlation for the six domains) and validity among several samples of women with sexual difficulties (Rosen et al., 2000; Meston, 2003; Wiegel, Meston & Rosen, 2005).
Changes in sexual distress from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Both partners will complete the Female Sexual Distress Scale, a 12-item measure designed to assess sexually related personal distress. Although designed for women, items are gender non-specific and could pertain to both women and men. Thus, no adaptations are required for use with male partners. This measure has demonstrated high internal consistency, test-retest reliability, discriminate validity, and construct validity (Derogatis et al., 2002).
Changes in Ambivalence over Emotional Expression from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Both partners will complete the Ambivalence over Emotional Expression Questionnaire (AEQ; King & Emmons, 1990). This measure assesses various aspects of ambivalence over expressing emotions (e.g., wanting to express but being unable to, expressing but not wanting to, or expressing and then regretting the decision). This self-report measure consists of 28 items. The AEQ has been shown to have good psychometric properties, including good internal stability, test-retest reliability and convergent validity (King & Emmons, 1990).
Changes in Dyadic Sexual Communication from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Dyadic sexual communication will be measured using the Dyadic Sexual Communication Scale (Catania, 1986). This measure is a 13-item scale that assesses partners' perceptions of their communication processes around sexual problems. Both members of the couple will complete this measure, which has demonstrated good reliability and a uni-factorial structure (Catania, Pollack, McDermott, Qualls, & Cole, 1990).
Changes in male sexual function from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Male partners will complete the International Index of Erectile Function (IIEF; Rosen, Riley, Wagner, Osterloh, Kirkpatrick & Mishra, 1997). The IIEF is a well-known instrument for assessing erectile function in men. It is comprised of 15 items, and 3 items to assess pelvic pain in men have been added to this measure, and these items are complimentary to those that appear in the FSFI.
Changes in self-compassion from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Both women and partners will complete the Self-Compassion Scale (Neff, 2003), a 26-item self-report inventory that assesses three different aspects of self-compassion.
Changes in experience of genito-pelvic pain from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  The Experience of Genito-Pelvic Pain Scale is comprised of 24 items focusing on the thoughts and feelings associated with pain during sexual activity. These include how the pain is experienced in relation to a romantic/sexual partner, how it affects one's sense of being a woman, and how it may generate negative emotions such as guilt and shame. This self-report measure is in the initial stages of development and will be partially validated during the course of the study. We expect that it will be sensitive to treatment changes. This measure will be completed by women only, given it focuses on pain during sexual activity.
Changes in experience of emotion regulation from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Emotion regulation will be measured in both partners using the Difficulties in Emotion Regulation Scale (DERS). The DERS is a brief, 36-item, self-report questionnaire designed to assess multiple aspects of emotion dysregulation. The DERS has been shown to have good psychometric properties, including good internal stability (α =0.93) and test-retest reliability. (Gratz & Roemer, 2004).
Changes in experience of compassionate love for partner from baseline to post-treatment, and 6-months post-treatment | Baseline, Post-treatment (12 weeks), and 6-months post-treatment (9 months from baseline)
  Both partners will complete a Compassionate love for partner scale, the specific close other version of the Compassionate Love scale (Sprecher & Fehr, 2005). Compassionate love is an attitude "containing feelings, cognitions, and behaviors that are focused on caring, concern, tenderness, and an orientation toward supporting, helping, and understanding the other, particularly when the other is perceived to be suffering or in need." The 21 items of this self-report inventory are rated on a scale from 1 (not at all true) to 7 (very true). Higher score indicates more compassionate love for the partner. Cronbach's alpha for this version of the scale was .94 (Sprecher & Fehr, 2005).

OTHER OUTCOMES:
History of trauma | Baseline
  Trauma, a potential moderator of treatment response, will be assessed using the Childhood Trauma Questionnaire (CTQ), a 28-item self-report measure focusing on emotional, physical, and sexual abuse, as well as physical and emotional neglect in childhood (Berstein et al., 2003). The CTQ is the only self-report measure of childhood victimization with demonstrated criterion validity to detect actual abuse and neglect histories. Scores range from 5 to 25 for each type of abuse and a total severity scale can also be computed.
Therapeutic alliance over the course of treatment | Treatment weeks 1, 4, 8, and 12
  Therapeutic alliance is defined by the expectations, agreements, and bond that forms between the therapist and the couple, as well between the therapist and each member of the couple (Pinsof & Caherall). We will measure this construct using the Revised Short Form Integrative Psychotherapy Alliance Scale for Couples, or the Couple Therapeutic Alliance Scale (CTASr-SF; Pinsof, Zinbarg, & Knobloch-Fedders, 2008) at four time points: at sessions 1, 4, 8, and 12. The CTASr-SF is a 12-item, self-report questionnaire. This scale is widely used in clinical work and research with couples, and alphas for all subscales is good (alpha = 0.70 or better). We have added a thirteenth item to assess ongoing satisfaction throughout the therapy process.
Treatment expectancies | Measured following randomization but before treatment begins
  Using visual analog scales, we will ask participants to rate their expectancies related to their beliefs of efficacy pertaining to the treatment to which they were randomized. This measure has been successfully used in our previous clinical trial research.
History of relationship conflict | Baseline
  Select questions from the Conflict Tactics Scale (CTS; Straus, Hamby, Boney-McCoy & Sugarman, 1996), and the NorVold Abuse Questionnaire (Swahnberg & Wijma, 2003) will be used to assess the presence of current (and past) physical and emotional abuse. These two measures were developed to assess the presence and history of relationship abuse (physical and emotional).
History of hormonal contraception use | Baseline
  A detailed question about the use of past and current contraceptives during the pre-treatment evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Bergeron, PhD, Principal Investigator — Université de Montréal; Natalie O Rosen, PhD, Principal Investigator — Dalhousie University
Locations (2):
- Canada (2):
  - Dalhousie University, Halifax, Nova Scotia
  - University of Montreal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Santerre-Baillargeon M, Rosen NO, Vaillancourt-Morel MP, Corsini-Munt S, Steben M, Mayrand MH, Bergeron S. Mediators of change in cognitive-behavioral couple therapy for genito-pelvic pain: Results of a randomized clinical trial. Health Psychol. 2023 Mar;42(3):161-171. doi: 10.1037/hea0001274. PMID 36862472
- [Derived] Corsini-Munt S, Bergeron S, Rosen NO, Steben M, Mayrand MH, Delisle I, McDuff P, Aerts L, Santerre-Baillargeon M. A comparison of cognitive-behavioral couple therapy and lidocaine in the treatment of provoked vestibulodynia: study protocol for a randomized clinical trial. Trials. 2014 Dec 23;15:506. doi: 10.1186/1745-6215-15-506. PMID 25540035